CLINICAL TRIAL: NCT03116854
Title: Real-world Use and Prognosis of Beta Blocker in Patients With Acute Coronary Syndrome in the Central China：a Prospective, Multicenter, Observational Research
Brief Title: Real-world Use and Prognosis of Beta Blocker in Patients With Acute Coronary Syndrome in the Central China
Acronym: UPB-ACS
Status: Completed | Type: Observational
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Principal Investigator, Chuanyu Gao, Director, Henan Institute of Cardiovascular Epidemiology
Other Study IDs: HenanICE201701
Record Dates: First submitted 2017-04-12; First posted 2017-04-17 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome; Beta Blockers; Prognosis
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Beta Blocker therapy is a mainstay of treatment following acute coronary syndromes (ACS), particularly acute myocardial infarction (MI). Studies have repeatedly demonstrated the benefit of Beta blocker therapy following either ST-segment elevation myocardial infarction (STEMI) or non-ST-segment elevation ACS,and Beta blocker therapy has been a performance measure used to grade hospital performance by the Centers for Medicare and Medicaid Services and Joint Commission on Accreditation of Healthcare Organizations.Although the benefit of Beta blocker therapy has been clearly demonstrated, the doses that have been used in many of these studies are significantly higher than those typically used currently in clinical practice.The benefit of Beta blockers has been ascribed to dose-related heart rate reduction,although alternative mechanisms for their benefit have also been proposed.In addition, the classical Beta blocker trials were performed decades ago, before the modern therapeutic era,which includes reperfusion therapy, potent antithrombotics, and statins. This raises the question of whether titration of Beta blocker therapy to the high doses that had been previously studied provides substantial incremental benefit in current clinical practice over the more frequently prescribed and clinically tolerated doses of Beta blockers.Moreover, a recent study has reported that high-dose Beta blockers were not superior to low-dose Beta blockers,aprovocative finding requiring validation. And until now, there has been no registry on patients with ACS about Between Beta-blocker Treatment in Henan, the most populated (about 100 million) and predominantly rural (66%)province in central China.

This multicenter, prospective, observational study is aimed to analyze the application status and long-term prognostic beneﬁt of beta-blockers in patients with acute coronary syndrome.

DETAILED DESCRIPTION:
1. Henan institute of cardiology epidemiology is responsible for design, data quality control and statistical analysis.
2. Data were collected using a uniformed Case Report Form(CRF) by trained staff at each hospital.
3. Sample size estimation: Based on retrospective observational cohort of ACS patients, 1-year mortality in beta-blocker recipients and non-beta-blocker recipients were 2.5% and 5.6%, respectively. To achieve a precision of 5% with an α of 0.05, the loss ratio of following-up is 15%.The investigators would need a sample of 3000.
4. Statistical analysis plan: the investigators will report summary statistics for patient characteristics, comorbidities, treatment strategies and outcomes. the investigators will also undertake the following prespecified subgroup analyses: age, sex, STE-ACS or NSTE-ACS, history of diabetes, history of hypertension, smoking.and analyze the association Between Beta-blocker Treatment and Long-term Mortality.
5. Quality assurance plan 1)Diagnosis of ACS is according to the third universal definition.2)Before registry, a training program on study objectives, data collection, and ACS management is given to the primary investigator and related staff at each participating center.3)Henan institute of cardiology epidemiology will regularly monitored at least 10% of CRFs for accuracy against medical records. If the CRFs are not completed with 98% accuracy, all CRFs are considered unqualified and this staff will be retrained.4)Before entering into the computer, data is queried for invalid and illogical values by research staff in Henan institute of cardiology epidemiology. Participating centres who has the high error rate of data, and no change in 6 months shall be deemed abandoned automatically; participating centres who has the high quality of data will be issued a certificate to reward.5)Investigator meeting will be annually held to conclude the progress, solve existing problems and strengthen program training.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years.
2. Patients with clinical evidence of acute coronary syndrome, including ST segment elevation myocardial infarction (STEMI), non ST segment elevation myocardial infarction (NSTEMI) and unstable angina.
3. Informed consent signed by patients or legal guardians.

Exclusion Criteria:

* Expected survival <12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anticipated 40 eligible sites in Henan province will participate. Each site will enroll patients who meet the inclusion criteria consecutively.
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-04-26 (Actual); Study Completion 2020-04-26 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular and cerebrovascular events | 1 year
  including all-caused death, nonfatal- myocardial infarction,and stroke

SECONDARY OUTCOMES:
Major adverse cardiovascular and cerebrovascular events | At discharge(an average of 10 days),6 month
  including all-caused death, nonfatal- myocardial infarction,and stroke
Coronary revascularization | 6 month,1 year
  including PCI,CABG,and PTCA
Re-hospitalized | 6 month,1 year
  Including hospitalization due to heart disease and noncardiac disease
Bleeding | At discharge(an average of 10 days),6 month,1 year
  according to GUSTO bleeding grade(excluding hemorrhage stroke)
Recurrent angina | At discharge(an average of 10 days)
  Recurrent angina during hospitalization
the aggravation of Angina pectoris | 6 month,1 year
  Angina pectoris graded of CCS(CanadianCardiovascularSociety) rating at least one level
New arrhythmia | At discharge(an average of 10 days)，6 month,1 year
  including atrial fibrillation，thoracicoutletsyndrome，ventricular fibrillation，sick sinus syndrome，grade atrioventricular block and so on

CONTACTS AND LOCATIONS:
Locations (1):
- Henan province people's hospital, Zhengzhou, Henan, China